CLINICAL TRIAL: NCT06939270
Title: Phase I/II Clinical Trial of CD73/AXL Targeted HypoSti.CAR-T Cells in Treating Patients With CD73/AXL Positive Advanced/Metastatic Solid Tumors
Brief Title: CD73/AXL Targeted HypoSti.CAR-T Cells in CD73/AXL Positive Advanced/Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-095
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor
Keywords: CD73/AXL; hypoxia; CAR-T Cells
MeSH Terms: conditions — Hypoxia | interventions — Albumin-Bound Paclitaxel; Injections; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD73/AXL.HypoSti.CAR-T cells (Experimental): Enrolled participants will be given a preconditioning regimen consisted of albumin-bound paclitaxel, cyclophosphamide and fludarabine before the infusion of CD73/AXL.HypoSti.CAR-T cells.
  Enrolled patients in this arm will be administered CD73/AXL.HypoSti.CAR-T cells in "3+3" based escalation manner.
  Interventions: Biological: CD73/AXL.HypoSti.CAR-T cells; Drug: Albumin-Bound Paclitaxel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: CD73/AXL.HypoSti.CAR-T cells — Dose escalation: Dose1 (1×10^6 cells/kg) , Dose 2(3×10^6 cells/kg) ,Dose 3 (1×10^7cells/kg); Dose expansion: RP2D.
Drug: Albumin-Bound Paclitaxel — Administered intravenously at dose of 100-200mg/m2 on day -5 .
  Other Names: Albumin-bound paclitaxel for Injection
Drug: Cyclophosphamide — Administered intravenously at a total dose of 15-30mg/kg on day -3 and day -2 .
  Other Names: Cyclophosphamide for Injection
Drug: Fludarabine — Administered intravenously at dose of 30mg/m2/d on day -3 and day -2.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
In this single-center, single-arm,prospective, open-label, phase 1/2 study, the safety and efficacy of novel autologous hypoxia-activated CAR-T cell therapy targeting CD73 and AXL ( CD73/AXL.HypoSti.CAR-T) will be evaluated in patients with CD73/AXL antigen positive advanced/metastatic solid tumors. In this clinical trial, at least 12 eligible patients in dose escalation period will be enrolled to receive 3 doses Of CD73/AXL.HypoSti.CAR-T cell therapy according to the "3+3" principle. In dose expansion period, additional at most 21 eligible patients will be enrolled to receive CD73/AXL.HypoSti.CAR-T cell therapy at dose of recommended phase 2 dose(RP2D).

DETAILED DESCRIPTION:
Currently, CAR T-cell therapy still faces significant challenges in its application to solid tumors due to multiple obstacles, including the lack of tumor-specific antigens, the complex immunosuppressive tumor microenvironment (TME), tumor heterogeneity, and on targeted/non-targeted (OTOT) toxicity. Previous studies have found that intratumoral hypoxic microenvironment facilitated the development and metastasis of tumor cells. Meanwhile, cytotoxic T cells, including CAR-T cells, struggle to survive and proliferate in this low-oxygen microenvironment.

CD73 (also known as 5'-nucleotidase) and AXL (a receptor tyrosine kinase) are both overexpressed in multiple solid tumors, but less so in normal tissues. They are both involved in regulating tumorigenesis, development, metastasis processes, correlating with inferior prognosis.Dual targeting of CD73 and AXL can effectively address antigen escape and tumor heterogeneity, representing a promising novel immunotherapy strategy.

In this study, combining hypoxia-activated precision with dual-targeting synergy,Investigators have developed a novel CD73/AXL.HypoSti.CAR-T that could effectively expand and survive in hypoxic TME ,offering enhanced efficacy and safety for solid tumors in animal models. Further clinical development is warranted to validate these promising preclinical results. So we conduct this clinical trial in order to test the the safety profiles and anti-tumor activities of CD73/AXL.HypoSti.CAR-T cell in vivo. In dose escalation period, at least 12 eligible patients will be enrolled and receive 3 doses of CD73/AXL.HypoSti.CAR-T cell therapy (1 × 10^6 cells/ kg, 3 × 10^6 cells/kg, 1 × 10^7 cells/kg) according to the "3+3" principle. In dose expansion period, additional at most 21 eligible patients will be enrolled to receive CD73/AXL.HypoSti.CAR-T cell infusion at RP2D, which is determined by data from dose escalation period, including occurrence of dose limiting toxicities (DLT), pharmacokinetics/pharmacodynamics, efficacy and other parameters, to furtherly evaluate the safety and efficacy profiles of CD73/AXL.HypoSti.CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (inclusive).
2. The Eastern Cooperative Oncology Group (ECOG) score ≤2 and Estimated life expectancy of more than 3 months.
3. Histopathological confirmed advanced or metastatic solid tumors failed to at least first-line treatment or initially diagnosed advanced/metastatic solid tumors that have no National Comprehensive Cancer Network (NCCN) guideline recommended standard firstline therapy. Tumor types include but are not limited to:biliary malignancies, pancreatic cancer, lung cancer, breast cancer, head and neck malignancies, gynecological tumors, etc.
4. The expression of CD73 or AXL antigen is≥50%.
5. At least one measurable lesion at baseline per RECIST version 1.1.
6. Fresh solid tumor samples or formalin-fixed paraffin embedded tumor archival samples within 6 months are necessary; Fresh tumor samples are preferred. Subjects are willing to accept tumor rebiopsy in the process of this study.
7. Adequate organ function as defined by the following criteria:

   * Absolute neutrophil count (ANC) ≥ 1 x 10^9/L, Platelet count ≥75 x 10^9/ L, hemoglobin (Hgb) ≥ 90g/L ;
   * Serum creatinine≤1.5 upper limit of normal (ULN) or creatinine clearance (as estimated by Cockcroft Gault) ≥60 mL/min;
   * Serum aspartate amino transferase (AST) and alanine aminotransferase (ALT), ≤3.0 x ULN (≤5 x ULN for patients with liver cancer or metastases); Total serum bilirubin ≤1.5 x ULN(≤3 x ULN for patients with liver cancer or metastases);
   * Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings;
   * International Normalized Ratio (INR) ≤ 1.5 times the upper limit of normal (ULN), and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN;
   * Baseline oxygen saturation >91% on room air.
8. Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to <= grade 1 toxicity (except for hematological toxicities and clinically non-significant toxicities such as alopecia).
9. Pregnancy tests for women of childbearing age shall be negative; Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
10. Ability to understand and sign a written informed consent document.

Exclusion Criteria:

1. Subjects are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
2. Received cytotoxic chemicals, monoclonal antibodies, immunotherapy, targeted therapy or other anti-tumor therapy within 4 weeks or 5 half-lives before enrollment.
3. Pregnant, lactating, or breastfeeding females.
4. Known positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS);Active infection of hepatitis B virus (HBV), or hepatitis C virus (HCV).
5. History of allergy or intolerance to study drug components.
6. Prior organ allograft transplantations or allogeneic hematopoietic stem cell transplantation.
7. Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
8. Known brain metastases or active central nervous system (CNS).Subjects with CNS metastases who were treated with radiotherapy for at least 3 months prior to enrollment, have no central nervous symptoms and are off corticosteroids, are eligible for enrollment, but require a brain MRI screening.
9. Previous or concurrent cancer within 5 years prior to treatment start except for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors.
10. Uncontrolled intercurrent illness, including ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
11. Active bleeding or known hemorrhagic tendency.
12. Vaccination within 30 days of study enrollment.
13. Being participating any other trials or withdraw within 4 weeks.
14. Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of treatment related adverse events (TRAEs). | Up to 12 months
  TRAEs are defined as any medical events since the initiation of CD73/AXL.HypoSti.CAR-T cell therapy . Cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) will be evaluated according to the standards released by American Society for Transplantation and Cellular Therapy (ASTCT) criteria in 2019, and the others will be graded by common terminology criteria for adverse events (CTCAE) V5.0.
Phase 1:Incidence of dose limiting toxicities (DLTs). | Up to 28 days after infusion.
  DLTs are defined as CD73/AXL.HypoSti.CAR-T cell therapy related adverse events within the first 28 days that meet the following criteria:
  * Grade 4 CRS or grade 3 CRS that is not resolved to grade 2 or lower within 2 weeks;
  * Grade 3 ICANS lasting for ≥7 days or Grade 4 ICANS;
  * Any other Grade ≥4 and Grade 3 AEs related to the CD73/AXL.HypoSti.CAR-T infusion that lasts for ≥14 days, except hematology toxicity.
Phase 1: RP2D | Up to 12 months.
  The recommended dose for phase 2 was determined through phase 1 study.
Phase 2: Objective response rate (ORR) . | Up to 3 years.
  ORR includes complete response(CR) and partial response (PR), as defined by investigators according to investigators Response Evaluation Criteria in Solid Tumours 1.1 (RECIST 1.1) or Immune Response Evaluation Criteria in Solid Tumours (iRECIST) criteria.

SECONDARY OUTCOMES:
Phase 1 and phase 2: Pharmacokinetics:Number and copy number of CD73/AXL.HypoSti.CAR-T cells . | Up to 12 months.
  Number and copy number of CD73/AXL.HypoSti.CAR-T cells were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (until CD73/AXL.HypoSti.CAR-T cells were not detected for two consecutive times) to detect the number and copy number of CD73/AXL.HypoSti.CAR-T cells, and to evaluate the pharmacokinetics of CD73/AXL.HypoSti.CAR-T.
Phase 1 and phase 2: Pharmacodynamics: Peak level of cytokines in serum. | Up to 28 days after infusion.
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP), ferritin. Peak was defined as the maximum post-baseline level of the cytokine.
Phase 2:Progression Free Survival (PFS) | Up to 3 years.
  PFS is defined as the time from the initiation of CD73/AXL.HypoSti.CAR-T cell therapy to documented disease progression or death.
Phase 2:Time to response (TTR). | Up to 3 years.
  TTR is defined as the time from the initiation of CD73/AXL.HypoSti.CAR-T cell therapy to first assessed CR or PR by investigators according to RECIST 1.1or iRECIST criteria.
Phase 2:Duration of response (DOR) . | Up to 3 years.
  DOR is defined as the time from objective response until documented tumor progression among responders.
Phase 2:Overall Survival (OS) | Up to 3 years.
  OS is defined as the time from the initiation of CD73/AXL.HypoSti.CAR-T cell therapy to documented disease progression or death.

OTHER OUTCOMES:
Relationship between infusion dose of CD73/AXL.HypoSti.CAR-T and efficacy. | Up to 12 months.
  The relationship between the number of CD73/AXL.HypoSti.CAR-T, copy number, cytokines level, and anti-tumor effect of CD73/AXL.HypoSti.CAR-T cells was analyzed. Peripheral blood was collected at the day of infusion (day 0), day1,day 4, day 7, day 11, day 14, day 28, at least once every month after 28 days, at least once every three months after half a year, and at least once every six months after a year. The number of CD73/AXL.HypoSti.CAR-T cells was detected by flow cytometry, and the copy number was detected by quantitative PCR (qPCR).
Dynamics characteristic of CD73/AXL.HypoSti.CAR-T cells and key molecular and cellular mechanisms of tumor resistance in vivo after infusion. | Up to 12 months.
  The dynamic changes of the number and copy number of CAR-T cells in patients after CD73/AXL.HypoSti.CAR-T treatment were analyzed. The peak, expansion pattern,continuous expansion time and evolution of CD73/AXL.HypoSti.CAR-T cells in vivo was summarized. To analyze the evolution of CD73/AXL antigen and other changes at the cellular or molecular level after treatment, and to summarize the key cellular and molecular mechanisms of resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital; Jianqing Xu, Ph.D, Study Director — Institutes of Biomedical Sciences, Fudan University
Locations (1):
- Biotherapeutic Department, Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No